CLINICAL TRIAL: NCT02732756
Title: Cognitive and Behavioral Effects of Sleep Restriction in Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CIN_ADHDsleep_001
Record Dates: First submitted 2016-03-24; First posted 2016-04-11 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Sleep; Attention; Adolescence
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep Restriction (Experimental): The Sleep Restriction condition will allow 6.5 hours in bed, which in previous research results in an average of 6.1-6.3 hours of nightly sleep. This condition reflects a realistic dose of sleep restriction (similar to the school-night sleep of 15-20% of healthy adolescents) that has been shown to be feasible and to induce daytime sleepiness, inattention, and irritability/moodiness in typically developing adolescents.
  Interventions: Behavioral: Shortened Sleep Duration
- Sleep Extension (Experimental): The Sleep Extension condition will allow adolescents to obtain 9 hours of nightly sleep (9.5 hours in bed, leaving up to ½ hour to fall asleep), which (a) is how long adolescents sleep during controlled trials of sleep satiation and naturally on non-school nights, (b) has been shown to result in a well-rested state, and (c) matches clinical recommendations for adolescents.
  Interventions: Behavioral: Healthy Sleep Duration

INTERVENTIONS:
Behavioral: Healthy Sleep Duration — This study examines healthy sleep duration as related to improved functioning in adolescents with ADHD. Adolescent participants will be instructed to go to bed at a time such that they are able to obtain 9 hours of nightly sleep (9.5 hours in bed, leaving up to ½ hour to fall asleep). Researchers will work with the adolescent and their family to problem-solve how to accomplish this sleep duration goal.
  Arms: Sleep Extension
Behavioral: Shortened Sleep Duration — This study examines shortened sleep duration as related to poorer functioning in adolescents with ADHD. Adolescent participants will be instructed to go to bed at a time such that they are in bed for 6.5 hours per night. Researchers will work with the adolescent and their family to problem-solve how to accomplish this sleep duration goal.
  Arms: Sleep Restriction

SUMMARY:
Adolescents with attention-deficit/hyperactivity disorder (ADHD) obtain less sleep than their typically developing peers. Observational studies indicate that inadequate sleep is correlated with impairment in adolescents with ADHD, but it remains unknown if sleep is causally related to impairment. This study will use an experimental sleep restriction and extension protocol to evaluate sleep as a contributor to clinically significant impairment and possible target for intervention in adolescents with ADHD.

DETAILED DESCRIPTION:
Teens with attention-deficit/hyperactivity disorder (ADHD) obtain less sleep than their peers, with up to 75% of youth with ADHD obtaining insufficient sleep. This is noteworthy since insufficient sleep is associated with a multitude of negative outcomes in typically developing teens, including academic underachievement, emotion dysregulation, and mental health problems - all outcomes that occur at higher rates among teens with ADHD. Our pilot work demonstrates that insufficient sleep is correlated with depression, behavior problems, and academic impairment in teens with ADHD specifically and insufficient sleep is clearly associated with greater attentional problems in typical teens. However, no experimental study has examined whether sleep duration is causally linked to attentional, behavioral, emotional, and academic impairments in teens diagnosed with ADHD. If sleep problems contribute to functional impairments in teens with ADHD, then they represent an overlooked treatment target. Experimental studies provide the strongest test of causality, and studies using at-home sleep restriction protocols in teens without ADHD show a causal link between shortened sleep duration and impairment. However, administering an at-home sleep restriction protocol may be especially challenging for teens with ADHD due to their difficulties with organizing bedtime and wake activities, as well as differences from healthy teens in biological circadian preference. Thus, a critical first step in examining sleep as causally related to impairment in teens with ADHD is documenting the feasibility of using an at-home sleep restriction protocol with this population. This study will (1) evaluate the feasibility of using an at-home sleep restriction protocol in teens with ADHD, and (2) collect preliminary data examining whether shortened sleep duration is causally linked to attentional, behavioral, emotional, and academic impairment in teens with ADHD. These goals will be accomplished by recruiting 54 teens with ADHD who will undergo a three-week sleep manipulation protocol. Specifically, a cross-over design will be used that includes a week of typical sleep followed by weeks of sleep restriction or sleep extension. Sleep functioning will be assessed during these three weeks with daily sleep diary and objective sleep measurement (i.e., actigraphy). After each sleep condition, teens and their parents will complete subjective and objective measures of attention, behavior, mood, and academics. Findings from this study will allow us to identify and address barriers to administering an at-home sleep restriction and extension protocol to teens with ADHD and pursue larger-scale experimental research examining sleep problems as causally linked to impairment. This research is clinically significant since teens with ADHD frequently experience a range of impairments that extend well into adulthood. If short sleep duration contributes to functional impairments in teens with ADHD, then sleep represents a modifiable and overlooked treatment target.

ELIGIBILITY:
Inclusion Criteria:

* Between 14 and 17 years of age.
* Estimated IQ ≥ 70.
* Meet full DSM-5 criteria for ADHD.
* Sufficient English language ability necessary to complete study measures.
* If applicable, the family must be willing to discontinue any treatment with a psychostimulant medication during the three-week sleep manipulation protocol.

Exclusion Criteria:

* Children with an autism spectrum disorder or diagnosed with psychosis, bipolar disorder, or obsessive-compulsive disorder based on the K-SADS diagnostic interview will be excluded.
* Children taking any psychiatric medication that is not a psychostimulant.
* Significant visual, hearing, or speech impairment.
* Organic brain injury or history of seizures.
* Symptoms of obstructive sleep apnea (OSA), periodic limb movement disorder (PLMD), or delayed sleep phase syndrome (DSPS).
* Obligations that require bedtime later than 10pm or waking prior to 5:30am any morning of the study.
* Daily consumption of >1 coffee or "energy drink" or >3 caffeinated sodas.
* Highly atypical sleep, defined as <6 hours or >9.5 hours on school nights per parent and adolescent report.
* Inability or refusal to refrain from automobile driving or other high-risk tasks that require vigilance during the sleep restriction week of the study.
* Finally, at the visit following the baseline week (week 1) of the sleep protocol, we will exclude teens whose actigraphs reflect an inability to consistently arise within 1 hour of the agreed-upon time.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Change in sleep duration | Following each of the two arms that each last one week.
  Sleep duration will be assessed with actigraphy for five days during each sleep restriction/extension experimental arm. The sleep duration outcome will be assessed as the change in average nightly sleep duration between the sleep restriction and sleep extension arms.

SECONDARY OUTCOMES:
Change in ADHD symptoms | Following each of the two arms that each last one week.
  ADHD symptoms will be assessed using parent and adolescent ratings at the end of each five-day period following each sleep restriction (Week A) and sleep extension (Week B) experimental arm. The ADHD symptom outcome will be assessed as the change in ADHD symptoms between the two week-long experimental arms.
Change in internalizing symptoms | Following each of the two arms that each last one week.
  Internalizing symptoms will be assessed using parent and adolescent ratings at the end of each five-day period following each sleep restriction (Week A) and sleep extension (Week B) experimental arm. The internalizing outcome will be assessed as the change in internalizing symptoms between the two week-long experimental arms.
Change in behavioral functioning | Following each of the two arms that each last one week.
  Oppositional symptoms will be assessed using parent ratings at the end of each five-day period following each sleep restriction (Week A) and sleep extension (Week B) experimental arm. The oppositional behavior outcome will be assessed as the change in oppositional behaviors between the two week-long experimental arms.
Change in cognitive functioning | Following each of the two arms that each last one week.
  Cognitive functioning will be assessed using neuropsychological test performance at the end of each five-day period following each sleep restriction (Week A) and sleep extension (Week B) experimental arm. The outcome will be assessed as the change in neuropsychological test performance between the two week-long experimental arms.
Change in emotion regulation | Following each of the two arms that each last one week.
  Emotion regulation will be assessed using parent and adolescent ratings at the end of each five-day period following each sleep restriction (Week A) and sleep extension (Week B) experimental arm. The emotion regulation outcome will be assessed as the change in emotion regulation between the two week-long experimental arms.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Becker SP, Epstein JN, Tamm L, Tilford AA, Tischner CM, Isaacson PA, Simon JO, Beebe DW. Shortened Sleep Duration Causes Sleepiness, Inattention, and Oppositionality in Adolescents With Attention-Deficit/Hyperactivity Disorder: Findings From a Crossover Sleep Restriction/Extension Study. J Am Acad Child Adolesc Psychiatry. 2019 Apr;58(4):433-442. doi: 10.1016/j.jaac.2018.09.439. Epub 2018 Nov 2. PMID 30768404